CLINICAL TRIAL: NCT05156775
Title: The Efficacy of Ultrasound-Guided Rhomboid Intercostal Block Versus Serratus Plane Block in Patients Undergoing Modified Radical Mastectomy: A Prospective Randomized Controlled Study.
Brief Title: The Efficacy of Ultrasound-Guided Rhomboid Intercostal Block Versus Serratus Plane Block in Mastectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Hamdy Alhassanin, Resident of Anesthesia, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34981/10/21
Record Dates: First submitted 2021-11-27; First posted 2021-12-14 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Mastectomy; Rhomboid Intercostal Block; Serratus Plane Block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous analgesia group (No Intervention): 35 Patients will receive intravenous morphine (mg) analgesia only.
- Serratus Plane Block (SPB) group (Experimental): 35 Patients will receive ipsilateral serratus plane block using 30 ml bupivacaine 0.25% at the level of the 5th rib.
  Interventions: Other: Serratus Plane Block (SPB)
- Rhomboid intercostal nerve block (RIB) group (Experimental): 35 Patients will receive ipsilateral rhomboid intercostal nerve block using 30 ml bupivacaine 0.25%.
  Interventions: Other: Rhomboid intercostal nerve block (RIB)

INTERVENTIONS:
Other: Serratus Plane Block (SPB) — While the patient is in the supine position, the arm will be abducted, the ultrasound probe will be placed over the mid-clavicular region of the thoracic cage in sagittal plane. Ribs will be counted until the fifth rib will be identified in the midaxillary line. the latissimus dorsi (superficial and posterior ), teres major (superior), and serratus muscle (deep and inferior)will be identified overlying the fifth rib. As an extra reference point, thoracodorsal artery will be used, this aids in the identification of the plane superficial to the serratus muscle, 30 ml 0.25 %bupivacaine will be injected between latissimus dorsi and serratus anterior muscles at the level of the 5th rib in the mid axillary line.
  Arms: Serratus Plane Block (SPB) group
Other: Rhomboid intercostal nerve block (RIB) — In the rhomboid intercostal nerve block (RIB) group, the patient will be placed in a lateral position with the affected breast at the top. The ipsilateral arm will be extended to the same level as the ipsilateral chest and breast, and the scapula will be moved outward. On the oblique sagittal plane, a high frequency (6-12MHz) linear ultrasound probe will be placed on the medial edge of the scapula. The US landmarks, trapezius muscle, rhomboid muscle, intercostal muscles, pleura, and lung will be identified. Under the aseptic condition, a 22-gauge needle will be inserted in the plan to the US probe at T5 to T6 levels. Then, 0.25% bupivacaine (30 mL) will be injected into the inter-fascial plane between the rhomboid major muscle and the intercostal muscle, the diffusion of bupivacaine in the fascia between the rhomboid muscle and the intercostal muscle will be visualized. Then, the patient will be positioned in supine position.
  Arms: Rhomboid intercostal nerve block (RIB) group

SUMMARY:
The aim of this study is to evaluate analgesic efficacy of ultrasound-guided rhomboid plane block or serratus plane block versus Intravenous opioid in patients undergoing modified radical mastectomy.

DETAILED DESCRIPTION:
Breast cancer is the most frequently diagnosed malignancy and is the leading cause of cancer-related death among the female population.

Modified radical mastectomy (MRM) is the standard surgical treatment for cancer breast, which is usually associated with moderate to severe acute postoperative pain. Adequate postoperative pain relief is important to improve functional outcomes and to accelerate recovery and decrease hospital stay.

The postoperative pain may last >3 to 6 months after surgery and may proceed to chronic pain, with an incidence of 20% to 30%. Because chronic pain has many negative effects on patients, it may decrease the overall quality of life and may be a potential source of chronic opioid use. Therefore, preventing chronic pain is essential in these patients. In this regard, good acute postoperative pain management strategies have a very important role.

Regional anesthesia techniques can provide good postoperative pain management and may cause less incidence of chronic pain.

Many analgesic techniques have been proposed to relieve acute postoperative pain, including intercostal block, local anesthetic (LA) infiltration, block, paravertebral block, serratus plane block (SPB), and rhomboid intercostal block (RIB) to relieve acute postoperative pain

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Scheduled for unilateral modified radical mastectomy.
* Age 18-65 years
* American Society of Anesthesiologists (ASA) physical status I- II

Exclusion Criteria:

* Patient refusal
* Coagulation disorders
* Body mass index > 35 kg/m2
* Uncooperative or psychiatric patients
* Infection at the injection site
* Patients with a history of allergy to local anesthetics
* Patients with a history of treatment for chronic pain
* Previous history of breast surgery or other chest surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-29 (Estimated); Study Completion 2022-05-29 (Estimated)

PRIMARY OUTCOMES:
The total rescue morphine (mg) consumption in the first 24 post-operative hours. | 24 hours postoperative
  Rescue analgesia in the form of 3 mg intravenous morphine (mg) will be given if the visual analog scale is ≥ 4 repeated with 10 minutes lockout interval till the visual analog scale becomes less than 3 guided with the occurrence of complications as nausea, vomiting, and respiratory depression.

SECONDARY OUTCOMES:
Post-operative pain assessed by visual analog scale (VAS) | 24 hours Postoperative
  Postoperative pain will be assessed using a visual analog scale after 15 minutes after admission to the Post-anesthesia care unit and, 2, 4, 6, 8, 12,16, and 24 hours postoperatively.
  VAS ranged from 0 to 10 (the lowest is less pain)
Heart rate | Intraoperative
  Heart rate (beats/min) will be recorded at baseline before induction, after induction, and before skin incision then every 15 minutes till the end of the operation
Mean arterial blood pressure | Intraoperative
  Mean arterial blood pressure will be recorded at baseline before induction, after induction, and before skin incision then every 15 minutes till the end of the operation
Time to first rescue analgesic request (minutes) | 24 hours Postoperative
  Time to the first rescue analgesic request (minutes) will be also recorded. Rescue analgesia in the form of 3 mg intravenous morphine (mg) will be given if the visual analog scale is ≥ 4
Intraoperative fentanyl consumption (µg). | Intraoperative
  Inadequate analgesia in the form of increase of heart rate or mean arterial blood pressure ≥ 20% above the baseline will be managed using 1µg/ kg of IV fentanyl. The total intravenous fentanyl consumption will be recorded at the end of the operation
Adverse effects | intraoperative or 24 hours Postoperative
  Any intraoperative or postoperative complications such as nausea, vomiting, hematoma, hypotension (defined as any decrease in mean arterial blood pressure of >20% of the preoperative baseline value), Bradycardia (defined as a decrease in heart rate < 50 beat/min), or pneumothorax will be recorded. Bradycardia will be treated by atropine intravenous injection (0.01 mg/kg) which may be repeated if needed. Hypotension will be treated by250 ml intravenous saline, and a bolus dose of intravenous Ephedrine 5 mg, which may be repeated if no response.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The supporting data will be available upon a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: One year after the end of the study